CLINICAL TRIAL: NCT05977920
Title: Fasciculations in Healthy Adults After Consumption of Caffeine: an Ultrasound Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zurich Regional Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-02103
Record Dates: First submitted 2023-05-21; First posted 2023-08-07 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Neurologic Symptoms
MeSH Terms: conditions — Neurologic Manifestations | interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: There is only one group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Only one Arm (Other): s. description
  Interventions: Other: Caffeine

INTERVENTIONS:
Other: Caffeine — s. description

SUMMARY:
Fasciculations are clinically defined as spontaneous intermittent contractions of a portion of muscles. Depending on associated symptoms they may be a sign of lower motor neuron disorder. The aim of this study is to investigate if fasciculations also occur in muscles after caffeine consumption and if there is a difference between the muscles of the arms and legs.

The primary endpoint is detecting fasciculations in the muscles of the arms and legs after the consumption of caffeine in healthy adults (20-35 years old and 35-50 years old) Secondary endpoints of the study compares the proportions of fasciculations between two age groups (20-35 years old and 35-50 years. A population of 26 subject per group and a total of 52 subject will be recruited for the study. A sample size of 26 in each group will have 90% power to detect a difference between the two groups using a Fisher's exact test with a 0.05 two-sided significance level.

Study Intervention Study participants will consume caffeine (6mg per kilogram bodyweight) before the second ultrasound screening.

Using ultrasound the sternocleidomastoideus, biceps brachii, interosseus dorsalis, quadriceps femoris, gastrocnemius and abductor hallucis will be measure for 120 seconds 1o minutes before and 45 minutes after caffeine consumption.

Study Duration and Schedule Estimated duration for the study will be around 6 months.

DETAILED DESCRIPTION:
Fasciculations are clinically defined as spontaneous intermittent contractions of a portion of muscles [8]. They can also be assessed with electromyography and are classified as a result of spontaneous depolarization of a lower motor neuron leading to the synchronous contraction of all of the skeletal muscle fibers within a single motor unit [9]. On ultrasound examination fasciculations are classified as involuntary twitching of small parts of the muscle, lasting for 0.2 - 1.0 seconds [10]. They result from spontaneous discharges of motor nerves, but the etiology and the site of origin of these discharges remains still uncertain and is controversially discussed [11, 12]. Depending on the associated symptoms they may be a sign of lower motor neuron disorder. They are a hallmark of amyotrophic lateral sclerosis, a neurodegenerative disease affecting upper motor neurons in the brain and lower motor neurons in the spinal cord, especially when they are widespread [13, 14]. Fasciculations can also be a normal phenomenon that almost everyone has experienced occasionally in their lives or more frequently in healthy subjects after exercise [15]. It is controversially discussed if fasciculations above the knee should raise the suspicion of a disorder even if there are no other signs of lower motor neuron affection. In a recent Dutch study the prevalence and distribution of fasciculations in healthy adults was assessed with ultrasound and it could be shown, that strenuous physical exercise causes a temporary increase in fasciculations but only in lower leg muscles in healthy adults [14]. However the fasciculations were screened only for 10 seconds 30 minutes after exercise. It is well known that the observation time for fasciculations should be 2 minutes to decide if a muscle is "fasciculation-free" [15]. The aim of this study is to investigate if fasciculations also occur in muscles after caffeine consumption and if there is a difference between the muscles of the arms and legs.

3 STUDY OBJECTIVES AND DESIGN 3.1 Hypothesis and primary objective The hypothesis about the primary endpoint, the comparison of two proportions, can be examined by a Fisher exact test.

The null hypothesis of the primary endpoint is, that there is no difference in the proportions of fasciculations below and above the knee.

The alternative hypothesis of the primary endpoint states a difference in the proportions of fasciculations below and above the knee.

Secondary objective / endpoint:

Secondary endpoints of the study compares the proportions of fasciculations between two age groupes (20-35 years old and 35-50 years old):

The hypothesis of the secondary endpoints are examined again by a Fisher exact test.

The null and alternative hypothesis of the secondary endpoints are analogous. 3.2 Primary and secondary endpoints The primary endpoint is detecting fasciculations in the muscles of the arms and legs after the consumption of caffeine in healthy adults (20-35 years old and 35-50 years old) 3.3 Study design Monocentric Cross-sectional study. 3.4. Study intervention See 4.3 Study procedures 4 STUDY POPULATION AND STUDY PROCEDURES 4.1 Inclusion and exclusion criteria, justification of study population A population of 26 subject per group and a total of 52 subject will be recruited for the study.

List the study inclusion criteria:

* Healthy subjects (male/female)
* Age 20-50 years old

List the study exclusion criteria:

* neurological symptoms
* any neurological disease including neuropathies, myopathies or radiculopathies in personal history
* systemic disease including vasculitis in personal history
* abnormal pulse in the arteria dorsalis pedis
* abnormal strength, sensation and tendon reflexes
* muscular atrophy in the studied muscles.

4.2 Recruitment, screening and informed consent procedure Recruitment will be done within our social circle and patient population. The investigators ask friends and acquaintances if they would like to take part in the study. If the investigators don't find enough test subjects in this way, the investigators will put up a notice at the University of Zurich or advertise online. The subjects who agree to participate in the study will be informed about the exact course of the study in a conversation and can then decide whether they agree to participate. Only when they have decided to participate in the study, the inclusion and exclusion criteria are queried on the basis of a precise anamnesis. This is followed by a neurological examination (sensitivity test, examination for paresis, cranial nerve status, reflexes, vibration sensation, standing and gait tests) as well as a measurement of blood pressure and pulse.

4.3 Study procedures

The planned overall study duration, including recruitment period will be 6 months. The recruitment and intervention will take place over 4 months. On the day of the examination, the subjects should appear rested (not overtired) and feel good. First, the blood pressure and pulse are measured. The neurological examination is carried out during the clarification of the inclusion and exclusion criteria after the anamnesis interview (see 4.2). The subjects should have taken at least 12 hours before the examination no caffeine and alcohol as well as drugs or medications. They should eat and drink normally and should not be sober. 10 minutes before taking caffeine, the ultrasound examination of the muscles is performed. The test subject is lying down during this procedure while being calm and relaxed without tensing their muscles. They should not be talking during both ultrasound examinations. Caffeine is taken in the form of coffee. It does not matter in the study whether they are regular coffee drinkers or not. Blood pressure and pulse are measured every 30 minutes after taking the caffeine for 2 hours. In total, the test takes 3 hours.

Using ultrasonography the sternocleidomastoideus, biceps brachii, interosseus dorsalis, quadriceps femoris, gastrocnemius and abductor hallucis will be measured for 120 seconds (with video recording) 10 minutes before and 45 minutes after caffeine consumption (6 mg per kilogram body weight).

4.4 Withdrawal and discontinuation In accordance with the Declaration of Helsinki a subject has the right to withdraw from the study at any time without giving reason. Subjects who are withdrawn by the Investigator because of an unacceptable adverse event will be termed a withdrawal" and will not be replaced. Under these circumstances the Investigator will institute the appropriate follow-up investigations in accordance with accepted standards of medical care including performance of tests at the time of withdrawal. Subjects who withdraw from the study for any reasons will not be replaced.

5 STATISTICS AND METHODOLOGY 5.1. Statistical analysis plan and sample size calculation

Methods:

For a comparison of the proportions of fasciculations above and below the knee a Fisher's exact test for a comparison of proportions is applied, using the R function [16] fe.ssize from the R package clinfun [17]. The investigators need to make assumptions about the following quantities:

* Significance level α. The investigators set α = 0.05.
* Assumed proportions: In the first group (fasciculations above knee), one expects p1 ∈ {0.6, 0.55}.

Note that for values of p1 close to 0 the number of patients needed varies substantially for small changes in p1. The investigators compute sample sizes for assumed group 2 proportions (fasciculations below knee) of p2 ∈ {0.1, 0.15}.

• Power, the probability of rejecting the null hypothesis of equal proportions in the two groups when the true difference is at least as assumed. The investigators compute sample sizes for power 1 - β ∈ {0.8, 0.9}.

Sample Size:

In Table 1 the investigators provide sample sizes for the above assumptions.

Significance level α Power 1 - β p1 p2 n per group for Fisher's exact test 0.05 0.05 0.05 0.05 0.8 0.8 0.8 0.8 0.6 0.6 0.55 0.55 0.1 0.15 0.1 0.15 17 22 19 25 0.05 0.05 0.05 0.05 0.9 0.9 0.9 0.9 0.6 0.6 0.55 0.55 0.1 0.15 0.1 0.15 20 26 24 32 Total number in study for Fisher's exact test 34 44 38 50 40 52 48 64

Table 1: Sample sizes.

A sample size of 26 in each group will have 90% power to detect a difference between proportions of p1 = 0.6 (fasciculations above knee) and p2 = 0.15 (fasciculations below knee) using a Fisher's exact test with a 0.05 two-sided significance level. This results in a total sample size of 52.

5.2. Handling of missing data and drop-outs The number of fasciculations can be viewed again, because the ultrasound examinations are recorded as a film and can be viewed again at any time. If data should nevertheless be lost, the relevant subject will be asked whether he can take part again on another day or whether new participants will be recruited.

Drop-outs are replaced by recruitment of new subjects. 6 REGULATORY ASPECTS AND SAFETY 6.1 Local regulations / Declaration of Helsinki This study is conducted in compliance with the protocol, the current version of the Declaration of Helsinki, the ICH-GCP, the HRA as well as other locally relevant legal and regulatory requirements.

6.2 (Serious) Adverse Events and notification of safety and protective measures An Adverse Event (AE) is any untoward medical occurrence in a patient or a clinical investigation subject which does not necessarily have a causal relationship with the trial procedure. An AE can therefore be any unfavourable or unintended finding, symptom, or disease temporally associated with a trial procedure, whether or not related to it.

A Serious Adverse Event (SAE) (ClinO, Art. 63) is any untoward medical occurrence that

* Results in death or is life-threatening,
* Requires in-patient hospitalisation or prolongation of existing hospitalisation,
* Results in persistent or significant disability or incapacity, or
* Causes a congenital anomaly or birth defect

Both Investigator and Sponsor-Investigator make a causality assessment of the event to the trial intervention, (see table below based on the terms given in ICH E2A guidelines). Any event assessed as possibly, probably or definitely related is classified as related to the trial intervention.

Relationship Description Definitely Temporal relationship Improvement after dechallenge* Recurrence after rechallenge (or other proof of drug cause) Probably Temporal relationship Improvement after dechallenge No other cause evident Possibly Temporal relationship Other cause possible Unlikely Any assessable reaction that does not fulfil the above conditions Not related Causal relationship can be ruled out

*Improvement after dechallenge only taken into consideration, if applicable to reaction

Both Investigator and Sponsor-Investigator make a severity assessment of the event as mild, moderate or severe. Mild means the complication is tolerable, moderate means it interferes with daily activities and severe means it renders daily activities impossible.

Reporting of SAEs (see ClinO, Art. 63) All SAEs are documented and reported immediately (within a maximum of 24 hours) to the Sponsor-Investigator of the study.

If it cannot be excluded that the SAE occurring in Switzerland is attributable to the intervention under investigation, the Investigator reports it to the Ethics Committee via BASEC within 15 days.

Follow up of (Serious) Adverse Events Describe the follow up procedures of participants terminating the study with reported ongoing (S)AEs until resolution or stabilisation.

Notification of safety and protective measures (see ClinO, Art 62, b) If immediate safety and protective measures have to be taken during the conduct of the study, the investigator notifies the Ethics committee of these measures, and of the circumstances necessitating them, within 7 days.

6.3 (Periodic) safety reporting An annual safety report (ASR) is submitted once a year to the local Ethics Committee by the Investigator (ClinO, Art. 43 Abs 1).

6.4 Amendments Substantial changes to the study setup and study organization, the protocol and relevant study documents are submitted to the Ethics Committee for approval before implementation. Under emergency circumstances, deviations from the protocol to protect the rights, safety and well-being of human subjects may proceed without prior approval of the Ethics Committee. Such deviations shall be documented and reported to the Ethics Committee as soon as possible.

Substantial amendments are changes that affect the safety, health, rights and obligations of participants, changes in the protocol that affect study objective(s) or central research topic, changes of study site(s) or of study leader and sponsor (ClinO, Art. 29).

A list of substantial changes is also available on www.swissethics.ch. A list of all non-substantial amendments will be submitted once a year to the competent EC together with the ASR.

6.5 Notification and reporting upon completion, discontinuation or interruption of the study Upon regular study completion, the Ethics Committee is notified via BASEC within 90 days (ClinO, Art. 38).

Provide a statement that the Sponsor-Investigator and any other competent authority may terminate the study prematurely according to certain circumstances, e.g:

The Sponsor-Investigator may terminate the study prematurely according to certain circumstances, e.g.

* Ethical concerns,
* Insufficient participant recruitment,
* When the safety of the participants is doubtful or at risk (e.g. when the benefit-risk assessment is no longer positive),
* Alterations in accepted clinical practice that make the continuation of the study unwise, or
* Early evidence of harm or benefit of the experimental intervention

Upon premature study termination or study interruption, the Ethics Committee is notified via BASEC within 15 days (ClinO, Art. 38).

6.6 Insurance In the event of study-related damage or injuries, the liability of the institution (Spital Wetzikon) provides compensation, except for claims that arise from misconduct or gross negligence.

ELIGIBILITY:
Inclusion criteria:

* Healthy subjects (male/female)
* age 20-50 years old

Exclusion criteria:

* Clinical neurological symptoms
* Clinical signs for Neuropathy
* Clinical signs for Myopathy
* Clinical signs for Vasculitis
* Clinical signs for heart disease
* Clinical signs for gastric or duodenal ulcera
* Any medicine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is detecting fasciculations in the muscles of the arms and legs after the consumption of coffein in healthy adults (20-35 years old and 35-50 years old) | 1 year
  We use ultrasound to detect the number of fasciculations before and after the consumption of caffeine in 6 muscles (arms and legs) to ascertain whether or not caffeine has an effect on the number fasciculations and if the muscles of either the upper or lower extremities are more involved. More details are provided in the detailed study description.

CONTACTS AND LOCATIONS:
Overall Officials: David Czell, Principal Investigator — Zurich Regional Health Center
Locations (1):
- GZO, Wetzikon, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No